CLINICAL TRIAL: NCT03837613
Title: Prognostic Value of Tumor Thickness of Buccal Mucosa Squamous Cell Carcinoma on the Incidence of Nodal Metastasis in the Neck: A Cohort Study
Brief Title: Prognostic Value of Tumor Thickness of Buccal Mucosa Squamous Cell Carcinoma on the Incidence of Nodal Metastasis.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mohamed Ghorab (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Mohamed Ghorab, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Other Study IDs: MohamedGhorabMSc
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Cancer; Squamous Cell Carcinoma
Keywords: cancer; squamous cell carcinoma; ultrasound; tumor thickness
MeSH Terms: conditions — Neoplasms; Carcinoma, Squamous Cell | interventions — Neck Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tumor tissue and the dissected cervical lymph nodes retained for histopathological study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (TT<4mm): Patients with a preoperative tumor thickness less than 4 mm. Intervention: tumor resection and neck dissection
  Interventions: Procedure: tumor resection and neck dissection
- Group 2 (TT >= 4mm): Patients with a preoperative tumor thickness equal to or more than 4 mm Intervention: tumor resection and neck dissection
  Interventions: Procedure: tumor resection and neck dissection

INTERVENTIONS:
Procedure: tumor resection and neck dissection — Surgical removal of the tumor with adequate safety margins. In addition to neck dissection to dissect the cervical lymph nodes.

SUMMARY:
Does the tumor thickness value of buccal squamous cell carcinomas, predict cervical nodal metastasis in clinically and radio-graphical neck negative (N0) thus sparing such patients unnecessary surgical procedures and it's associated morbidities? The aim of the study is to evaluate the prognostic value of tumor thickness cut off 4 mm in predicting cervical nodal metastases in a population of Egyptian patients presenting with Buccal Squamous Cell Carcinoma. The hypothesis is that patients with tumor thickness less than 4 mm will present with significantly less cervical nodal metastasis.

DETAILED DESCRIPTION:
Patients will be recruited from the outpatient clinics of Al Monofia university hospital, Cairo University Hospital and National Cancer Institute. Patients who fits the inclusion criteria and are motivated and consent to enter the study will be included. Patient recruitment will continue until the target sample size is reached.

Patients data will be collected including personal data, medical history, family history, and classification of the tumor according to the TNM classification system. Patients will be assessed preoperatively with a transcutaneous high frequency probe ultrasound to measure the maximal tumor thickness in millimeters using a 10MHz superficial probe and the lymph nodes in the neck region. In addition to clinical examination and palpation of the neck lymph nodes. Patients will then undergo tumor resection surgery with adequate safety margins under GA with nasotracheal intubation. Selective neck dissection will then be performed. The specimens will be submitted for histopathological examination.

Patients will receive standard post operative care based on the recommendation of the oncologist. Adjunct chemo or radiotherapy will be administered when deemed necessary. Wound care and dressings will be administered as needed.

Patients will be categorized into two groups based on the tumor thickness (exposure).

For the primary outcome, the data source will be the measurement of tumor depth based on Berslow method as discussed in the review of literature, obtained from ultrasonography and recorded in millimeters.Tumor width recorded in (mm) will also be obtained from the ultrasonography as it may be a source of confounders. Further, histological grade of the lesion will also be recorded.

Two confounding factors are highlighted and may be sources of bias and attempt to control for them in the statistical analyses will be made.

Appropriate statistical methods will be used after collection of the data and sources of confounders will be controlled for during analyses in subgroup An attempt to control for tumor width and histological grade in subgroup analyses

All data will be entered electronically. Patients' files are to be stored in numerical order and stored in secure and accessible place. All data will be maintained in storage for 1 year after completion of the study. Data monitoring committee is independent from the sponsor and competing interest.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian patients with BSCC (T all N0) not previously operated or treated with adjunctive therapy. They should present with no clinical signs of neck lymph nodes involvement.

Exclusion Criteria:

* Patients with lesions secondary to another primary site.
* Patients previously removed a primary oral surgery tumor in another site
* Patients with clinical or radiographic evidence of cervical nodal metastases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Egyptians Patients presenting to Cairo University dental Hospital, National Cancer Institute, and Al Monofia university hospital who fits the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Cervical nodal metastasis | one week after the surgery
  Number of patients with positive cervical nodal metastasis

SECONDARY OUTCOMES:
Tumor thickness | one week after the surgery
  Correlation between the tumor thickness measured preoperatively by ultrasound versus the tumor thickness measured from the histopathological specimen

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ghorab, BSD, Principal Investigator — Cairo University
Locations (1):
- Cairo University - Faculty of Oral and Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang SH, Hwang D, Lockwood G, Goldstein DP, O'Sullivan B. Predictive value of tumor thickness for cervical lymph-node involvement in squamous cell carcinoma of the oral cavity: a meta-analysis of reported studies. Cancer. 2009 Apr 1;115(7):1489-97. doi: 10.1002/cncr.24161. PMID 19197973
- [Background] Ota Y, Aoki T, Karakida K, Otsuru M, Kurabayashi H, Sasaki M, Nakamura N, Kajiwara H. Determination of deep surgical margin based on anatomical architecture for local control of squamous cell carcinoma of the buccal mucosa. Oral Oncol. 2009 Jul;45(7):605-9. doi: 10.1016/j.oraloncology.2008.08.010. Epub 2008 Nov 20. PMID 19026588
- [Background] Deshpande G, Das S. Tumor Thickness: A predictor of nodal disease in early squamous cell carcinomas of buccal mucosa. Gulf J Oncolog. 2015 May;1(18):37-43. PMID 26003104